CLINICAL TRIAL: NCT02821650
Title: Low-smoke Chulha in Indian Slums
Brief Title: A Study to Test the Impact of an Improved Chulha on Respiratory Health of Women and Children in Indian Slums
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of COVID-19, we could complete the follow-ups
Sponsor: Maastricht University (Other)
Responsible Party: Principal Investigator, Megha Thakur, External PhD student at CAPHRI school of public health and primary care, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 076-00051
Record Dates: First submitted 2016-06-21; First posted 2016-07-01 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Signs and Symptoms, Respiratory; Air Pollution, Indoor
MeSH Terms: conditions — Signs and Symptoms, Respiratory

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention arm will be administered with improved cook stoves (TEJ- Traditional stove to Efficient stove in Jhuggi).
  Interventions: Other: TEJ (Traditional stove to Efficient stove in Jhuggi)
- control (No Intervention): control arm will continue using traditional cook stoves (chulha) or a combination of the traditional stove and the kerosene/diesel stove.

INTERVENTIONS:
Other: TEJ (Traditional stove to Efficient stove in Jhuggi) — TEJ (means 'Bright' in Hindi) is an improved cook stove, locally designed and manufactured, aimed at reducing the indoor air emissions and improving health outcomes. 'Jhuggi' is a Hindi word which stands for a 'slum dwelling'
  Arms: Intervention

SUMMARY:
The present study documents a randomized controlled study investigating the efficacy of improved cookstove on the personal exposure to air pollution and the respiratory health of women and children in an Indian slum. The improved cookstove is based on co-creation of a low-smoke chulha with local communities in order to support adaption and sustained uptake. The study is conducted in notified and non-notified slums in Bangalore, India. The study design is be a 1:1 randomised controlled intervention trial. Outcomes include change in lung function (FEV1/FVC), incidence of pneumonia, change in personal PM2.5 and CO exposure, incidence of respiratory symptoms (cough, phlegm, wheeze and shortness of breath), prevalence of other related symptoms (headache and burning eyes), change in behaviour and adoption of the stove.

DETAILED DESCRIPTION:
Noting the significant health impact of the use of solid fuels and traditional cooking systems on (public) health indicators, it is imperative to find clean cooking solutions for urban slum dwelling communities. While several efforts have been made to reduce indoor air pollution in India, most efforts focused on "enhancing stove energy efficiency, and not reducing emissions." Also, use of a strict top-down approach in the community was responsible for many unsuccessful projects. The current project is based on principles of co-creation, involving the local community in designing and producing clean cook stoves; a more scalable and sustainable solution than fully subsidized efforts.

The aim of the present trial is to reduce the levels of household air pollution and improve the respiratory health of women and children by using a locally designed and manufactured improved cook stove. The study design will be a 1:1 randomised controlled intervention trial.

The intervention group will receive a locally designed and manufactured improved cookstove (low-smoke chulha). The control group will continue using the traditional cookstove (chulha) or a combination of the traditional stove and the kerosene/diesel stove.

The first part of project EXHALE was based upon an iterative process of co-creation of a low-smoke chulha with local communities in order to support adaption and sustained uptake. A qualitative study was conducted to gain insight into the cooking practices and challenges faced with the traditional stoves. Workshops were conducted where people were involved in creating an ideal stove, using thermocol blocks. Feedback was continuously used to optimize the design of the cookstove. Improved cookstoves were evaluated in a qualitative study in a slum called Siddhaarthanagar colony in Peenya, Bangalore.

Block randomization will be performed to reduce bias and achieve balance in the allocation of participants to treatment arms. Block sizes vary between two, four and six households to reduce the possibility of knowing the next randomization allocation. The study will be single-blinded (data-analyst). Randomization is stratified for having a child aged 5 years or younger or not.

Data for the questionnaires and for the assessment of pneumonia will be collected using a tablet computer with a pre-formatted questionnaire sheet. All data collection and storage devices will be password protected. Only supervisors and the main researcher will have access to the data files, identifiers, and keys. An intention-to-treat analysis will be conducted in order to ensure external validity of the study and minimize bias.

Since the intervention is not a clinical intervention, and does not have adverse effect on the participants, a data monitoring committee has not been formed. However, to review and keep track of the progress of the trial, a clinical advisory committee comprising of relevant experts has been formed.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥18 years who cooked more than 50% of the meals during the past 30 days (primary cook) and one child per household (0-5 years) will be included
* Both households with and without children will be included
* Women/mothers who are capable of being interviewed
* Will not migrate in the upcoming 2 months as far as the participants can predict
* Households cooking solely with traditional stove (chulha) or a combination of a traditional stove and a kerosene/diesel stove will be included

Exclusion Criteria:

* Households with a cooking area outside the house will be excluded
* Persons who are seriously ill will be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Lung function | 1 year
  Measure change in lung function (FEV1/FVC) as measured by spirometry in the primary cook
Pneumonia | 1 year
  Measure incidence of pneumonia for children ≤5 years. The incidence of pneumonia for children ≤5 years will be determined according to the definition of the WHO Integrated Management of Childhood Illness (IMCI). Screening for pneumonia will be done every three months for one year

SECONDARY OUTCOMES:
PM2.5 and CO exposure | 1 year
  Personal exposure to PM2.5 and CO will be measured for the primary cook using personal samplers
Respiratory symptoms | 1 year
  Measure incidence of respiratory symptoms, including cough, phlegm, wheeze and shortness of breath for the primary cook
Other related symptoms | 1 year
  Measure prevalence of other related symptoms, including headache and burning eyes for the primary cook

CONTACTS AND LOCATIONS:
Overall Officials: Constant Paul Van Schayck, PhD, Principal Investigator — Maastricht University, Caphri School of Public Health and Primary Care
Locations (4):
- India (4):
  - Ashrayanagar slum, Bangalore, Karnataka
  - Mathikere slum, Bangalore
  - Muneshwaranagar slum, Bangalore
  - Peenya slum, Bangalore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thakur M, Boudewijns EA, Babu GR, Winkens B, de Witte LP, Gruiskens J, Sushama P, Ghergu CT, van Schayck OCP. Low-smoke chulha in Indian slums: study protocol for a randomised controlled trial. BMC Public Health. 2017 May 16;17(1):454. doi: 10.1186/s12889-017-4369-6. PMID 28511647
- See also: Related Info — http://thorax.bmj.com/content/early/2018/06/20/thoraxjnl-2017-210952